CLINICAL TRIAL: NCT06497452
Title: A Prospective, Observational Study to Explore the Efficacy and Safety of Salvage Therapy With Glofitamab in a Real-world Setting in Chinese Adult Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma.
Brief Title: A Study of Efficacy and Safety of Glofitamab in Combination With Salvage Therapy in a Real-world Setting in Chinese Adult Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma.
Acronym: GLOFTST
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: GLOFTST
Record Dates: First submitted 2024-07-05; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: B-cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — glofitamab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational Cohort
  Interventions: Drug: Glofitamab

INTERVENTIONS:
Drug: Glofitamab — Glofitamab will be administered at the discretion of the physician per local clinical practice and local labeling

SUMMARY:
The purpose of this study is to assess the efficacy and safety in the real-world settings of glofitamab in combination with salvage therapy among Chinese adult patients with relapsed or refractory B-cell non-hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed as B-NHL
* Relapse or refractory to previous treatment
* Participants who will be treated with glofitamab

Exclusion Criteria:

* Participant who currently participates in or with plan to participate in any interventional clinical trial
* Any other reason that, in the investigator's opinion, makes the participant unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who will be treated with glofitamab (known as being recommended and having the intention to be treated with glofitamab at the time of signing informed consent) or have initiated glofitamab treatment within three months prior to enrollment and after the indication approval will be observed in this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Best Complete Response Rate (bCRR) Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | Baseline up to EOT (approximately 9 months)

SECONDARY OUTCOMES:
Best Overall Response Rate (bORR) Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | Baseline up to EOT (approximately 9 months)
Duration of Response (DoR) | From the date of the first occurrence of a documented CR or partial response (PR) to the date of progression, relapse, or death from any cause, whichever occurs first (up to approximately 24 months)
Duration of Complete Response (DoCR) | From the date of the first occurrence of a documented CR to the date of progression, relapse, or death from any cause, whichever occurs first (up to approximately 24 months)
PFS Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | Baseline up to end of study (approximately 24 months)
Event Free Survival (EFS) Assessed by Investigator per Lugano Response Criteria for Malignant Lymphoma | From the start of glofitamab treatment to any treatment failure including disease progression, relapse, initiation of new antilymphoma therapy (NALT), or death from any cause, which occurs first (up to approximately 24 months)
Overall Survival (OS) | From the start of glofitamab treatment until the date of death from any cause (up to approximately 24 months)
Time to Next Treatment (TTNT) | From the start of glofitamab treatment to the initiation of next-line treatment (up to approximately 24 months)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China